CLINICAL TRIAL: NCT03585881
Title: Evaluation of Accuracy of 3DPrinted Windowed Bracket- Positioning Guide Compared To Thermoformed Transfer Tray For Orthodontic Indirect Bonding A Randomized Controlled Trial
Brief Title: Accuracy of 3DPrinted Windowed Bracket- Positioning Guide Compared To Thermoformed Indirect Bonding Tray
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Ibrahim, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEBD-CU-2018-04-18
Record Dates: First submitted 2018-06-08; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Inaccurate Transfer and Bond Failure of Conventional Indirect Bonding Tray; Accuracy of Bracket Transfer and Bond Failure Rate of Digitally Printed Transfer Tray With Windows and Conventional Thermoformed Transfer Tray

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- window bracket positioning tray (Experimental)
  Interventions: Device: 3DPrinted Windowed Bracket- Positioning tray
- conventional indirect boning tray (No Intervention)

INTERVENTIONS:
Device: 3DPrinted Windowed Bracket- Positioning tray — 3 D printed tray with windows for accurate positioning of brackets
  Arms: window bracket positioning tray

SUMMARY:
this study was aimed to evaluate of accuracy of 3DPrinted windowed Bracket- Positioning Guide in compare to Thermoformed Transfer Tray For Orthodontic Indirect Bonding

ELIGIBILITY:
Inclusion Criteria:

1. Age: above 13 years.
2. Complete set of permanent teeth including second molar.
3. No sex predilection.
4. Class I Mild to moderate crowding (4-6 mm).

Exclusion Criteria:

1. Surface enamel defect that compromise bonding
2. No or poor patient's compliance.
3. Psychological problems.
4. Pathology at the site of intervention.
5. Insufficient crown height that contradicts bonding of brackets.
6. Labial and buccal Restorations.
7. Poor oral hygiene.
8. Severely rotated teeth

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of 3D printed transfer tray with windows& conventional thermoformed transfer tray | immediate
  using digital measurements on 3 shape software in mm degrees

SECONDARY OUTCOMES:
chairside time | immediate
  digital stopwatch in seconds
immediate bond failure | immediate
  counting after bonding number of brackets or tubes failed immediately